CLINICAL TRIAL: NCT02778698
Title: Compassionate Use of an Intravenous Fat Emulsion Comprised of Fish Oil in The Treatment of Parenteral Nutrition Induced Liver Injury in Children
Brief Title: Compassionate Use of Omegaven
Status: Approved for marketing | Type: Expanded Access
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Edward Everett DO, Principal Investigator, Geisinger Clinic
Other Study IDs: OMEGAVEN
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Cholestasis
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides

INTERVENTIONS:
Dietary Supplement: Omegaven

SUMMARY:
This expanded access protocol is for infants or children with conditions preventing them from taking in enough nutrients from food and must receive nutrition intravenously. Standard intravenous nutrition contains fat emulsion made from soybean. If this fat emulsion is given over a long period of time, it can cause problems within the liver and if persistent and not addressed can even lead to severe and/or permanent injury to the liver.

It is believed that a type of fish oil blend, called Omegaven®, may be used in place of the soybean fat blend. The Omegaven® fish oil blend may greatly reduce the risk of liver injury.

Omegaven® is not approved by the Food and Drug Administration (FDA). It is only offered under an "expanded access" protocol as an alternative to the soybean fat blend.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Older than 14 days and less than 5 years of age
3. Direct bilirubin value is greater than 2 mg/dL
4. Be expected to require intravenous nutrition for at least an additional 28 days
5. Parent/legal guardian has agreed to provide consent/parental permission

Exclusion Criteria:

1. Patients who have a congenitally lethal condition (e.g. Trisomy 13).
2. Patients who have clinically severe bleeding not able to be managed with routine measures.
3. Patients who have evidence of a viral hepatitis or primary liver disease as the primary etiology of their cholestasis.
4. Patients who have other health problems such that survival is extremely unlikely even if the infant's cholestasis improves.

5 The parent/legal guardian is unwilling to provide consent/parental permission.

Ages: 15 Days to 5 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Everett, DO, Principal Investigator — Geisinger Clinic